CLINICAL TRIAL: NCT05880212
Title: Implementation of the Specific Treatment of Problems of the Spine (STOPS) Approach in Bangladesh: a Prospective Sequential Comparison
Brief Title: Implementation of the Specific Treatment of Problems of the Spine Approach in Bangladesh
Acronym: STOPS-Bangla
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammad Ali (Other)
Collaborators: Hasna Hena Pain, Physiotherapy and Public Health Research Center (HPRC) (Unknown); La Trobe University (Other)
Responsible Party: Sponsor-Investigator, Mohammad Ali, PhD researcher, Uttara Adhunik Medical College
Organization: Uttara Adhunik Medical College (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HEC22334
Record Dates: First submitted 2023-05-04; First posted 2023-05-30 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Chronic Low-back Pain
Keywords: Chronic low back pain; Physiotherapy; Usual care; STOPS; Implementation trial; Bangladesh; Physiotherapist
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to the trial hypothesis and knowledge of the fact that two treatment options are being compared.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual physiotherapy care (Active Comparator): One physiotherapy assessment, 10 x 45-minute sessions of usual care physiotherapy (over a 10-week period), plus 1 x 45-minute followup session of usual care physiotherapy after 6 months.
  Interventions: Other: Usual physiotherapy care
- Individualized (STOPS) physiotherapy (Experimental): One physiotherapy assessment, 10 x 45-minute sessions of individualised (STOPS) physiotherapy (weekly for 10 weeks), plus 1 x 45-minute followup session of individualised (STOPS) physiotherapy after 6 months.
  Interventions: Other: Individualized (STOPS) physiotherapy

INTERVENTIONS:
Other: Usual physiotherapy care — In Phase 1, physiotherapists will provide treatment for participants with chronic low back pain in accordance with their current standard physiotherapy practice. Physiotherapists will be free to choose the treatment approach they wish to.
  Arms: Usual physiotherapy care
Other: Individualized (STOPS) physiotherapy — In Phase 3, participants will receive individualized physiotherapy in accordance with the Specific Treatment of Problems of the Spine (STOPS) approach modified for chronic low back pain. Treatment will be individualized on the basis of biopsychosocial assessment findings including dominant pain type (nociceptive, neuropathic or nociplastic), pathoanatomical subgroups (if any), and other barriers to recovery (eg. inflammation, depression, anxiety, stress, catastrophising, pain self-efficacy, and unhelpful motor control strategies). Available treatment strategies will include individualized education/advice, exercise, manual therapy, activity modification/facilitation, goal setting, motor control optimisation, cognitive-behavioural strategies, inflammation management, pain management strategies, sleep management, work management, and relaxation approaches.
  Arms: Individualized (STOPS) physiotherapy

SUMMARY:
The goal of this implementation trial is to evaluate the clinical outcomes associated with usual physiotherapy care compared to individualized physiotherapy in accordance with the Specific Treatment of Problems of the Spine (STOPS) approach in patients with chronic low back pain (CLBP). The main questions it aims to answer are:

* Is the STOPS approach more effective than usual care physiotherapy among patients with CLBP?
* Is STOPS physiotherapy cost-effective compared to usual physiotherapy care for patients with CLBP.
* Does STOPS training improve the quality of care among Bangladeshi physiotherapists?

DETAILED DESCRIPTION:
The goal of this implementation trial is to evaluate the clinical outcomes associated with usual physiotherapy care compared to individualized physiotherapy in accordance with the Specific Treatment of Problems of the Spine (STOPS) approach in patients with chronic low back pain (CLBP). The main questions it aims to answer are:

* Is the STOPS approach more effective than usual care physiotherapy among patients with CLBP?
* Is STOPS physiotherapy cost-effective compared to usual physiotherapy care for patients with CLBP.
* Does STOPS training improve the quality of care among Bangladeshi physiotherapists?

In phase I, patients with CLBP will be treated with usual physiotherapy care. In phase II, Bangladeshi physiotherapists will be provided with a STOPS training program by the Australian developers of STOPS. In phase III, the trained Bangladeshi physiotherapists will treat patients using the STOPS approach.

Clinical patient outcomes will be evaluated in Phase 1 and Phase 3 (pre and post implementation).

Physiotherapists' self-confidence and implementation behaviour will be evaluated before and after STOPS training.

A qualitative study of physiotherapists' and patients' experiences will be conducted after the completion of the usual care (Phase I) and STOPS treatment programs (Phase III).

ELIGIBILITY:
Inclusion Criteria:

Physiotherapists:

Qualified physiotherapists and physiotherapy assistants in Bangladesh who are involved in low back pain management and working in either or both trial settings will provide the treatment in phases 1 and 3. To be eligible, physiotherapists and physiotherapy assistants must be willing to participate in all phases of the trial (Phases I, II, and III). They must have completed the organised STOPS training course led by the original Australian developers (Jon Ford and Andrew Hahne), where the assessment and treatment protocols will be taught in Phase II.

Patients:

1. A primary complaint of either:

   1. low back pain, defined as pain between the inferior costal margin and the inferior gluteal fold with or without referral into the leg(s)

      or
   2. referred leg pain, defined as predominately unilateral posterior leg pain extending below the knee, or anterior thigh pain, with or without back pain
2. Duration of the current episode of primary complaint lasting for greater than 3 months (chronic stage of the injury)
3. Aged between 18 and 65 (inclusive)
4. Fluency in English or Bengali sufficient to complete questionnaires and to enable understanding of the intervention
5. Agreeing to refrain from other interventions wherever possible for the 10-week treatment period of the trial, aside from consultations with medical practitioners, medication, and any exercises already being undertaken

Exclusion Criteria:

Physiotherapist:

Not willing to participate in the study for all 3 phases.

Patient:

1. Red flag pathologies such as active cancer under current treatment, risk of spinal fracture, signs of potential infection, and major systemic inflammatory disease.
2. Signs of cauda equina syndrome based on bladder or bowel disturbance and/or imaging
3. Current pregnancy, or childbirth within the last 6 months, as this could impair the ability to undertake exercises, and could also cause back and leg symptoms that are not related to the subgroups under investigation
4. Spinal injections within the last 6 weeks, as we wish to study treatment effects independent of the effects of injections
5. Any history of lumbar spine surgery, as there is already considerable research evaluating the efficacy of post-surgical rehabilitation programs
6. A pain intensity score of less than 2/10 on the numerical pain rating scale due to low severity.
7. Minimal activity limitation, evidenced by a baseline ability to perform ALL of (walk, sit, and stand for one hour or more and no sleep disturbance at night), as we wish to exclude people with low severity.
8. Inability to walk safely, such as severe foot drop causing regular tripping, as the interventions in the trial include walking for most participants.
9. Planned absence of more than one week during the treatment period (such as holidays).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Activity limitation | Primary endpoint will be 26 weeks post-enrolment.
  Oswestry Disability Questionnaire (ODI). Measured from 0-100% with lower scores meaning less disability.
Back Pain Intensity | Primary endpoint will be 26 weeks post-enrolment.
  0-10 numerical pain rating scale, average over the previous week. Lower scores indicate a better outcome.
Leg Pain Intensity | Primary endpoint will be 26 weeks post-enrolment.
  0-10 numerical pain rating scale, average over the previous week. Lower scores indicate a better outcome.

SECONDARY OUTCOMES:
Work hours missed | 5, 10, and 26-weeks post enrolment
  Number of work/housework hours missed during the past 7 days (continuous scale from 0 to 50). Lower score indicated less hours missed (better outcome)
Work productivity | 5, 10, and 26-weeks post enrolment
  0-10 numerical rating scale of how much pain affected work productivity in the last 7 days. Score 0-10, with lower scores indicating less interference with work productivity.
Short-Form Örebro Musculoskeletal Pain Screening Questionnaire (ÖMPSQ-SF) | 5, 10, and 26-weeks post enrolment
  The total score ranges between 1 and 100, with higher scores indicating a worse outcome.
Health-related quality of life (EQ-5D-5L) | 5, 10, and 26-weeks post enrolment
  Utility scores will be calculated from the EuroQOL-5D-5L, with scores ranging from -0.148 to 0.949 (higher scores indicate better quality of life)
Depression, Anxiety and Stress Scales - DASS-21 | 5, 10, and 26-weeks post enrolment
  The DASS-21 measures symptoms of stress, anxiety and depression, with a total composite score ranging from 0-63 with higher scores indicating more severe symptoms of distress.
Pain Self Efficacy | 5, 10, and 26-weeks post enrolment
  Pain Self Efficacy Questionnaire (PSEQ). A raw score is presented with a range from 0 - 60, where high scores indicate greater levels of confidence in dealing with pain (better outcome).
Pain Catastrophizing | 5, 10, and 26-weeks post enrolment
  Pain Catastrophizing Scale (PCS). The score ranges from 0 to 52. A higher score denotes more catastrophizing (worse outcome)
Sleep quality | 5, 10, and 26-weeks post enrolment
  Insomnia Severity Index (ISI-7). Score ranges from 0 to 28, with higher scores indicating worse sleep quality (worse outcome)
Central Sensitisation symptoms | 5, 10, and 26-weeks post enrolment
  Central Sensitisation Inventory (CSI-9). Score ranges from 0 to 36, with higher scores indicating more symptoms indicative of potential central sensitisation
Inflammatory symptoms | 5, 10, and 26-weeks post enrolment
  The 4-item clinical inflammation score will measure low back-related inflammatory symptoms. Scores range from 0 to 4, with higher scores indicating more inflammatory symptoms (worse outcome)
Treatment Credibility | 5, 10, and 26-weeks post enrolment
  Treatment credibility questionnaire. Scored 0-10. A higher score indicates greater confidence in the treatment (better outcome).
Healthcare utilization | 5, 10, and 26-weeks post enrolment
  A patient diary will be used to track healthcare service utilization, imaging, and medication. These are recorded descriptively.
Participant adherence with treatment | 5, 10, and 26-weeks post enrolment
  Participant adherence with treatment will be determined via a self-administered 0-10 rating scale, with higher scores indicating greater adherence with treatment (better outcome).
Global rating of change | 5, 10, and 26-weeks post enrolment
  Global change will be measured on a 7-point scale ranging from "very much worse" to "very much better". Scores range from 1-7, with a higher score indicating greater improvement.
Satisfaction with treatment | 5, 10, and 26-weeks post enrolment
  Participants will rate their satisfaction with physiotherapy treatment on a 5-point Likert scale, with ratings from "very satisfied" to "very dissatisfied".
Adverse events | 5, 10, and 26-weeks post enrolment
  Adverse effects events (harmful or unpleasant) will be recorded descriptively in the therapists clinical notes.
Qualitative interviews | 10 weeks post-enrolment
  Semi-structured interviews relating to the patient's experiences with the Usual care and STOPS physiotherapy will be conducted.
Pain severity | 5, 10, and 26-weeks post enrolment
  Brief Pain Inventory. Average of the four pain severity items, scores range from 0-10, lower scores indicate less pain severity.
Pain interference | 5, 10, and 26-weeks post enrolment
  Brief Pain Inventory. Average of the seven pain interference items, scores range from 0-10, lower scores indicate less pain interference.
Back Pain Intensity | 5, 10 and 52-weeks post enrolment
  0-10 numerical pain rating scale, average over the previous week. Lower scores indicate a better outcome.
Leg Pain Intensity | 5, 10 and 52-weeks post enrolment
  0-10 numerical pain rating scale, average over the previous week. Lower scores indicate a better outcome.
Activity limitation | 5, 10 and 52-weeks post enrolment
  Oswestry Disability Questionnaire (ODI). Measured from 0-100% with lower scores meaning less disability.

OTHER OUTCOMES:
Physiotherapists' self-confidence in low back pain management | After 26 weeks of phases 1 and 3. After the completion of phase 2 training
  Practitioner Self-Confidence Scale. Scored 4-20 where higher scores indicate worse self-confidence towards clinical management of low back pain (worse outcome).
Physiotherapists' implementation behaviour | At the end treating the usual care group, and again at the end of treating the individualised (STOPS) physiotherapy group.
  Implementation behaviour questionnaire (DIBQ-t) will be used. The questionnaire includes 26 items, with each item rated on a 5-point Likert scale. A total score from 0-100 is derived, with higher scores indicate stronger implementation behaviours. (better outcome)
Physiotherapists' experiences | At the end treating the usual care group, and again at the end of treating the individualised (STOPS) physiotherapy group.
  Physiotherapists' experiences with implementing usual care and STOPS physiotherapy will be assessed via qualitative semi-structured interviews.
Treatment effect modifier: Pain type | Effect modifiers are measured at baseline, and their potential impact determined on outcomes at week 5, 10, and 26
  Pain type (categorised as nociceptive, neuropathic, or nociplastic dominant pain) is being pre-specified as a potential treatment effect modifier on the primary outcome measures. It is hypothesised that patients with neuropathic pain will derive additional benefit of STOPS physiotherapy over usual care.
Treatment effect modifier: Disability | Effect modifiers are measured at baseline, and their potential impact determined on primary outcomes at week 5, 10, and 26
  Disability (measured using the Oswestry Disability Questionnaire - score from 0-100%) is being pre-specified as a potential treatment effect modifier on the primary outcome measures. It is hypothesised that patients with higher disability scores will derive additional benefit from STOPS physiotherapy over usual care.
Treatment effect modifier: Prognosis (Orebro short-form screening questionnaire) | Effect modifiers are measured at baseline, and their potential impact determined on primary outcomes at week 5, 10, and 26
  Prognosis (measured on the 0-100 Orebro short-form) is being pre-specified as a potential treatment effect modifier on the primary outcome measures. It is hypothesised that patients with higher Orebro scores will derive additional benefit from STOPS physiotherapy over usual care.
Treatment effect modifier: Duration of symptoms | Effect modifiers are measured at baseline, and their potential impact determined on primary outcomes at week 5, 10, and 26
  Duration of symptoms (measured on a continuous scale in weeks) is being pre-specified as a potential treatment effect modifier on the primary outcome measures. It is hypothesised that patients with higher duration of symptoms will derive additional benefit from STOPS physiotherapy over usual care.
Mediator analysis: pain self-efficacy | Change in pain self-efficacy from baseline to 10 weeks and 26 weeks
  Mediator analyses will determine the potential mechanisms of action for the individualised (STOPS) physiotherapy, with the following potential mediator identified a-priori:
  Does pain self-efficacy (measured on the 0-60 pain self-efficacy scale) mediate the effect of individualised physiotherapy on primary outcomes
Mediator analysis: inflammatory symptoms | Change in clinical inflammation score from baseline to 10 weeks and 26 weeks
  Mediator analyses will determine the potential mechanisms of action for the individualised (STOPS) physiotherapy, with the following potential mediator identified a-priori:
  Does inflammation (measure on the 0-4 clinical inflammation scale) mediate the effect of individualised physiotherapy on primary outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Ali, MPhil, Principal Investigator — Uttara Adhunik Medical College Hospital
Locations (1):
- Uttara Adhunik Medical College Hospital, Dhaka, Uttara, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data collected during the trial will be available upon specific request t the researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 12 months of the study completion date
Access Criteria: Other researchers can request access to the data they require for a specific purpose. A data sharing agreement will need to be signed outlining the nature and restrictions on the use of the data for a specific purpose. Requests can be sent to the Investigators, or the La Trobe University Human Ethics Committee.

REFERENCES:
- [Derived] Ali M, Ford JJ, Hossain A, Danazumi MS, Hahne AJ. Implementing individualised physiotherapy using the Specific Treatment of Problems of the Spine (STOPS) approach for chronic low back pain in Bangladesh: Protocol for a prospective sequential comparison clinical trial. Contemp Clin Trials. 2025 Jul;154:107960. doi: 10.1016/j.cct.2025.107960. Epub 2025 May 21. PMID 40409680